CLINICAL TRIAL: NCT02492815
Title: An Observational Study to Evaluate the Effectiveness and Safety of Ipilimumab, Administered During the European Expanded Access Programme in Pretreated Patients With Advanced (Unresectable or Metastatic) Melanoma
Brief Title: PAN-EU Utilization, Effectiveness and Safety of Ipilimumab Administered in EAP Patients With Advanced Melanoma
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-367
Record Dates: First submitted 2015-06-03; First posted 2015-07-09 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Population with condition and without condition: Participating in EAP

SUMMARY:
Observational study to evaluate the effectiveness and safety of ipilimumab, administered during the European expanded access programme (EAP) in pretreated patients with advanced (unresectable or metastatic) melanoma.

DETAILED DESCRIPTION:
Minimum age: 18 years old (at time of inclusion in the CA184-367- but 16 for the EAP)

ELIGIBILITY:
Inclusion Criteria:

* Patients have been enrolled in the EAPs
* Patients still alive must provide informed consent if required by local regulations
* Deceased patients are eligible per local regulations, their legal representatives must provide informed consent if required by local regulations

Exclusion Criteria:

* There are no specific exclusion criteria in this observational study other than the exclusion criteria of the EAP

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients participating in Expanded Access Program
Sampling Method: Non-Probability Sample
Enrollment: 1773 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) of patients enrolled in the European ipilimumab EAP | Upto 60 month study period

SECONDARY OUTCOMES:
Demographic characteristics (age, weight, gender, race) of patients enrolled in the European ipilimumab EAP collected from medical charts | Upto 60 month study period
Clinical characteristics (biological values, stage of initial diagnosis, primary location of melanoma) of patients enrolled in the European ipilimumab EAP collected from medical charts | Upto 60 month study period
Frequency of discontinuing or skipping ipilimumab administrations among patients enrolled in the European ipilimumab EAP collected from medical charts | Upto 60 month study period
Reasons for discontinuing or skipping ipilimumab administrations among patients enrolled in the European ipilimumab EAP collected from medical charts | Upto 60 month study period
Treatment outcomes in specific sub-populations of patients enrolled in the European ipilimumab EAP collected from medical charts | Upto 60 month study period
Influence of demographic characteristics (age, weight, gender, race) on effectiveness and safety outcomes among patients enrolled in the European ipilimumab EAP collected from medical charts | Upto 60 month study period
Influence of clinical characteristics (biological values, stage of initial diagnosis, primary location of melanoma) on effectiveness and safety outcomes among patients enrolled in the European ipilimumab EAP collected from medical charts | Upto 60 month study period

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (2):
  - Local Institution, Boston, Massachusetts
  - Outcome Sciences Inc Dba Outcome, Boston, Massachusetts
- Local Institution, Linz, Austria
- Local Institution, Brussels, Belgium
- Local Institution, Prague, Czechia
- Local Institution, Odense C, Denmark
- Local Institution, Rouen, France
- Elbe Klinikum Buxtehude, Buxtehude, Germany
- Local Institution, Debrecen, Hungary
- Local Institution, Dublin, Ireland
- Local Institution, Napoli, Italy
- Local Institution, Amsterdam, Netherlands
- Local Institution, Oslo, Norway
- Local Institution, Moscow, Russia
- Local Institution, Valencia, Spain
- Local Institution, Zurich, Switzerland
- Local Institution, Guildford, Surrey, United Kingdom

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx